CLINICAL TRIAL: NCT05580575
Title: Evaluation of Wear Experience With Daily Disposable and Monthly Replacement Toric
Brief Title: Evaluation of Wear Experience With Daily Disposable and Monthly Replacement Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jennifer Fogt, PI, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022H0270
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Astigmatism Bilateral
Keywords: contact lenses; astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Daily disposable lens worn first, reusable lens worn second (Experimental): Subject will wear each contact lenses for 30 days during the day only.
  Interventions: Device: Daily disposable toric soft contact lens; Device: Monthly replacement toric daily wear soft contact lens
- Reusable lens worn first, daily disposable lens worn second (Experimental): Subject will wear each contact lenses for 30 days during the day only.
  Interventions: Device: Daily disposable toric soft contact lens; Device: Monthly replacement toric daily wear soft contact lens

INTERVENTIONS:
Device: Daily disposable toric soft contact lens — Daily disposable toric soft contact lens
Device: Monthly replacement toric daily wear soft contact lens — Monthly replacement toric daily wear soft contact lens

SUMMARY:
Comparison of wear experience with daily disposable and monthly replacement soft contact lenses in contact lens wearers who have astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be current soft lens wearers in both eyes.
* Subjects must have 20/25 or better distance visual acuity with current lenses (entering acuity).
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI)
* Ability to give informed consent
* Willing to spend time for the study. Subjects will be required to attend two study visits and wear contact lenses on days between study visits.
* Either gender
* Any racial or ethnic origin

Exclusion Criteria:

* Participants cannot be pregnant or lactating.
* Participants cannot be current wearers of the study lenses
* No current ocular inflammation or infection as assessed by the study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Complete Eye Care of Medina, Medina, Minnesota
  - The Ohio State University College of Optometry, Columbus, Ohio
  - ProCare Vision Center, Granville, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 4 screen failures at the first visit.
Groups:
- Daily Disposable Lens Worn First, Reusable Lens Worn Second (30 Days); Reusable Lens Worn First, Daily Disposable Lens Worn Second (30 Days): Subject will wear contact lenses for 30 days during the day only.
  Daily disposable toric soft contact lens: Daily disposable toric soft contact lens
  Monthly replacement toric daily wear soft contact lens: Monthly replacement toric daily wear soft contact lens
Period: Overall Study
Arm/Group | Daily Disposable Lens Worn First, Reusable Lens Worn Second (30 Days) | Reusable Lens Worn First, Daily Disposable Lens Worn Second (30 Days)
Started | 31 | 32
Completed | 28 | 31
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Daily Disposable Lens Worn First, Reusable Lens Worn Second; Reusable Lens Worn First, Daily Disposable Lens Worn Second: Subject will wear contact lenses for 30 days during the day only.
  Daily disposable toric soft contact lens: Daily disposable toric soft contact lens
  Monthly replacement toric daily wear soft contact lens: Monthly replacement toric daily wear soft contact lens
- Total: Total of all reporting groups
Arm/Group | Daily Disposable Lens Worn First, Reusable Lens Worn Second | Reusable Lens Worn First, Daily Disposable Lens Worn Second | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Categorical [Count of Participants; unit: Participants] — Population: Drop out subjects were not analyzed.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 28 | 31 | 59
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Drop out subjects not analyzed.
  years | 31 (10.8) | 31.9 (9.2) | 31.5 (10)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Drop out subjects not analyzed.
  Participants
    Female | 18 | 16 | 34
    Male | 10 | 12 | 22
    Transgender Female | 0 | 1 | 1
    Transgender Male | 0 | 1 | 1
    Nonbinary | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Drop out subject data not analyzed.
  Participants
    Hispanic or Latino | 2 | 4 | 6
    Not Hispanic or Latino | 25 | 27 | 52
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Drop out subjects not analyzed.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 4 | 2 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 22 | 24 | 46
    More than one race | 0 | 5 | 5
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Drop out subjects not analyzed.
  Participants
    United States | 28 | 31 | 59

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Survey of Overall Comfort
Description: Visual analog scale survey of comfort from 0 to 100, with 0 anchored as "poor" and 100 as "excellent"
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Daily Disposable Lens: Daily disposable toric soft contact lens: Daily disposable toric soft contact lens
- Reusable Lens: Monthly replacement toric daily wear soft contact lens: Monthly replacement toric daily wear soft contact lens
Arm/Group | Daily Disposable Lens | Reusable Lens
Number analyzed (Participants) | 59 | 59
units on a scale | 71.6 (26.3) | 63.2 (28.9)

ADVERSE EVENTS:
Time Frame: Entire study participation, about 60 days.
Arm/Group | Daily Disposable Lens | Reusable Lens
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/61
Other Adverse Events (participants affected / at risk) | 0/63 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT05580575/Prot_SAP_000.pdf